CLINICAL TRIAL: NCT05750680
Title: Interaction Between Direct Oral Anticoagulants and Drug-metabolizing Enzyme Inducers
Brief Title: DOCE Study Interaction Between Direct Oral Anticoagulants and Drug-metabolizing Enzyme Inducers
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, De Candia Erica, Prof.ssa Erica De Candia, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3981
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Thromboembolism, Venous
MeSH Terms: conditions — Atrial Fibrillation; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: DOACs — outpatients visited in anticoagulation clinics with a prescription of DOAC for atrial fibrillation and venous thromboembolism and concomitant antiepileptic drug will perform a blood draw for measurement of dabigatran, rivaroxaban, apixaban and edoxaban

SUMMARY:
Aim of the study is to investigate whether the influence of drugs inducing of CYP 3A4 isoenzyme of CYP450 and P-gp transporter significantly affect plasma levels of DOACs in patients with NVAF and venous thromboembolism

DETAILED DESCRIPTION:
Aim of the study is to investigate whether the influence of drugs inducing of CYP 3A4 isoenzyme of CYP450 and P-gp transporter significantly affect plasma levels of DOACs in patients with NVAF and venous thromboembolism. Also the difference between DOACs inducing both CYP3A4 and P-gp transporter (rivaroxaban and apixaban) and DOACs inducing the P-pg transporter only will be investigated. Thriomboembolic and bleeding events during the study duration will be registered and correlated to the measured DOAC plasma levels.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of nonvalvular atrial fibrillation or a diagnosis of venous thromboembolism who are taking direct oral anticoagulants according to current guidelines and concomitant enzyme inducers antiepileptic drugs; patients available for a 12 months follow up; patients who can sign informed consent

Exclusion Criteria:

* patients who stop antiepileptic drugs; age <18 yo patients not willing to perform blood draw or not available for a 12 months follow up; patients who cannot sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For sample size calculation we used data from a pilot study on 10 patients and controls. A significant difference of subject frequency with DOAC plasma concentrations below the expected peak value, respectively 35% and 10% for patients using or not using EI/AED, was defined as the primary end-point. A sample size of 40 subjects in each group was estimated for 80% power and alfa = 0.05
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
measurement of trough plasma levels of DOACs | 12 months
  measurement of trough plasma levels of DOACs in patients with NVAF and VTE under concomitant therapy with enzyme inducer antiepileptic drugs (EI-AED) and comparison with NVAF and VTE DOAC- treated patients with no EI-AED concomitant therapy

SECONDARY OUTCOMES:
measurement of peak plasma levels of DOACs in patients treated and not treated with EI-EAD | 12 months
  measurement of peak plasma levels of DOACs in patients treated and not treated with EI-EAD and registration of clinical outcomes of thromboembolic and bleeding events during the study duration

CONTACTS AND LOCATIONS:
Overall Officials: Erica De Candia, MD, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS Rome
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided